CLINICAL TRIAL: NCT07172815
Title: Evaluating the Safety and Efficacy of PDE-5 Inhibitor: Tadalafil as a Treatment for Early Stages of Alzheimer's Disease
Brief Title: PDE5 Inhibitor for Alzheimer's Disease
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 174242
Record Dates: First submitted 2025-08-29; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Alzheimer Disease
Keywords: Alzheimers; PDE5 Inhibitors; Blood Brain Barrier Dysfunction
MeSH Terms: conditions — Alzheimer Disease | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active drug: PDE5 inhibitor (Placebo Comparator)
  Interventions: Drug: tadalafil
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: tadalafil — Once daily dose of Tadalafil will be commenced at 10 mg for 2 weeks, followed by an increase to 20 mg for another 2 weeks and finally increased to 40 mg.
  Arms: Active drug: PDE5 inhibitor
Drug: Placebo — Matched Placebo will be taken once daily.
  Arms: Placebo

SUMMARY:
Alzheimer's disease is the most common cause of dementia in the elderly population. The disease is characterised by the presence of abnormal proteins in the brain, primarily β-amyloid (Aβ) and tau. Recent evidence suggests that Phosphodiesterase-5 (PDE-5) enzyme inhibitors may hold therapeutic promise in the treatment of early AD. Findings showed that daily low-dose tadalafil (a PDE5 inhibitor that can cross the BBB) administration in patients with erectile dysfunction and MCI increased relative regional cerebral blood flow in the postcentral gyrus, precuneus, and brainstem. However, the long-term effects of tadalafil on AD progression and biomarkers are not known. However, there is limited evidence regarding its safety and efficacy in AD patients. The primary objective of this study is to assess the safety and tolerability of long-term (1 year) tadalafil treatment in patients who are Aβ-positive MCI and early AD based on NIA-AA criteria. Additionally, the secondary objective of this study is to assess the change in cognitive performance from baseline to follow-up, evaluated using neuropsychometric testing, in MCI and AD patients who are undergoing treatment with tadalafil for 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving and capacity to give informed consent.
2. An individual who can act as a reliable study partner with regular contact.
3. Participants must meet the clinical criteria of MCI or AD.
4. Age from 50 years.
5. Mini-Mental State Examination (MMSE) score of 22-28.
6. Rosen Modified Hachinski Ischemic score ≤4.
7. Fluency in English and evidence of adequate premorbid intellectual functioning
8. Likely to be able to participate in all scheduled evaluations and complete all required tests.

Exclusion Criteria:

1. Any contraindications to the use of tadalafil.
2. Significant neurological disease other than MCI due to AD that may affect cognition.
3. MRI/CT showing unambiguous aetiological evidence of cerebrovascular disease.
4. Current presence of a clinically significant major psychiatric disorder.
5. Current clinically significant systemic illness that is likely to result in deterioration of the patient's condition or affect the patient's safety during the study.
6. Any previous enrolment in clinical trials within the last 3 months.
7. History of epilepsy, where seizures or treatment could have contributed to cognitive impairment.
8. ST Elevation Myocardial infarction within the last 1 year.
9. History of cancer within the last 5 years, except localised skin cancer.
10. Other clinically significant abnormality on physical, neurological or laboratory examination that could compromise the study or be detrimental to the patient.
11. History of alcohol or drug dependence or abuse within the last 2 years.
12. Current use of narcotic medications which could affect cognition.
13. Patients who have been involved in a monoclonal antibody study are excluded unless it is known that they were receiving placebo in that trial.
14. Women of childbearing potential.
15. Any contraindications to MRI scanning, including contraindications for the use of contrast agents, such as renal failure with the estimated glomerular filtration rate of less than 30 ml/minute or known allergy to gadolinium-based contrast agents.
16. Hypersensitivity to PDE-5 inhibitors.
17. Patients who are taking nitrates (see detailed list of nitrate medications in section 7.5).
18. Severe cardiac diseases.
19. Patients with unstable angina or angina occurring during exercise or patients with symptomatic coronary artery disease.
20. Patients with New York Heart Association Class 2 or greater heart failure in the last 6 months.
21. Patients with uncontrolled arrhythmias, hypotension (< 90/50 mmHg), or uncontrolled hypertension.
22. Patients with a stroke within the last 6 months.
23. Patients with pericardial constriction.
24. Patients with life-threatening arrhythmias.
25. Patients with severe renal impairment, defined by eGFR <30 mL/min/1.73 m² or the need for dialysis, and severe hepatic Impairment or any evidence of hepatic failure.
26. Any other contraindication listed in SmPC.
27. Patients who take one or more of the following medications: PDE-5 inhibitors other than tadalafil, any other investigational drugs other than tadalafil, potent inhibitors of CYP3A4 (see detailed list of drugs and consumables in section 7.5), any anti-amyloid or anti-tau therapies, any other investigational therapies for Alzheimer's disease, and any therapy that may affect Alzheimer's disease, as per the judgement of the Investigator.
28. [Only applicable for those agreeing to undertake an optional lumbar puncture] Any contraindications of lumbar puncture, including raised intracranial pressure (ICP) with suspected mass effect, skin infections at the puncture site, suspected spinal epidural abscesses, and cellulitis. Individuals with bleeding disorders that may increase the risk of bleeding (e.g. known bleeding diathesis, anticoagulant therapy, thrombocytopenia, abnormal coagulation parameters like prolonged Prothrombin Time (PT), prolonged activated Partial Thromboplastin Time (aPTT), and abnormal International Normalized Ratio (INR) will be excluded from having lumbar puncture.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
To assess the safety and tolerability of long-term (1 year) tadalafil treatment in MCI and early AD patients. | Data will be collected at screening, baseline, 3-month, 6-month, 9-month and 12-month follow-up.
  To assess the safety and tolerability of long-term (1 year) tadalafil treatment in MCI and early AD patients using composite outcome measure of the adverse events evaluated from the safety measurements.
  This will be assessed by the number of participants using a composite measure generated from abnormal vital signs, abnormal 12-lead ECG readings, abnormal laboratory (blood) tests, abnormal physical exam findings, and abnormal neurological/psychiatric evaluation.

SECONDARY OUTCOMES:
To assess the change in cognitive performance from baseline to follow-up evaluated using neuropsychometric testing (change in ADAS-Exec) in MCI and AD patients who are undergoing treatment with tadalafil for 1 year. | Neuropsychometric assessments will be collected at screening, baseline, 6 months and 12 months.
  Change in combined scores on neuropsychometric testing
  • ADAS-Exec Z score

IPD SHARING:
Plan to Share IPD: No